CLINICAL TRIAL: NCT03450642
Title: Complement Diagnosis of Acute Appendicitis
Acronym: CDAA
Status: Completed | Type: Observational
Sponsor: University of Exeter (Other)
Collaborators: Royal Devon and Exeter NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 1112/131544
Record Dates: First submitted 2015-08-05; First posted 2018-03-01 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Acute Appendicitis
MeSH Terms: conditions — Appendicitis | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation: Patients presenting with right Iliac Fosse pain
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Complement cascade components C3, C4, iC3b and TCC serum concentrations were measured over the time course from t= admission, 4,8,12,23,47,71 hours or until discharge.

SUMMARY:
Acute appendicitis is a common condition requiring urgent surgery but is often difficult to distinguish from other non-surgical conditions such as urinary infections, pelvic inflammatory disease and non-specific abdominal pain. Delay in diagnosis can result in significant morbidity and potential mortality. Currently, there is no one diagnostic test available and raised inflammatory markers such as C-reactive protein (CRP) and White Blood Count (WBC) along with an evolving clinical picture, help guide management. However, these markers are slow to respond to inflammation and are non-specific for appendicitis. The Complement cascade is an immune response to inflammation and infection involving three pathways which activate a number of proteins in the blood. Monitoring the absolute levels of these proteins should provide a faster and differential diagnostic test. The investigators propose a pilot trial to measure concentrations of Complement cascade activation biomarkers in the blood during hospital admissions for acute right lower abdominal pain, a symptom of appendicitis. Further, analysis of the differential Complement cascade pathway activation could potentially identify underlying pathology allowing the clinicians to target therapies.

DETAILED DESCRIPTION:
The proposed study is a pilot study on a cohort of participants recruited at emergency admission with acute right iliac fossa pain (right lower abdominal pain) to the Royal Devon & Exeter Hospital Accident & Emergency department. The pilot trial will collect one urine sample on admission and blood over a time course for each patient to record blood plasma levels of Complement proteins during hospital admissions with suspected appendicitis. The assay schedule is detailed in Table 1 below. The trial will perform additional Complement cascade activation tests on routine blood samples taken during the patient's stay in hospital. In addition 3 trial samples will be taken at time intervals that will capture the early Complement cascade response. Those patients going onto surgery will have a total of 5 additional trial samples taken, with 2 samples taken intra-operatively whilst under anaesthesia. From our previous experience in a similar pilot study CPOP (Complement cascade Predictors of Procedural Outcome), the investigators have introduced a blood taking 'curfew window' in which trial sample No. 2 & 3 must not take place between the hours of midnight and 0600 hrs. This is to incorporate the wishes of patients and improve compliance with the study. Sample analysis will be performed in parallel in the clinical chemistry laboratory for assays of CRP and the complement proteins C3 and C4. The additional trial assays will be performed by Prof Shaw's research post doctoral assistant in the clinical chemistry laboratory and in the Medical School. A fresh frozen urine sample will be acquired from the routine urine sample given on all admissions for RIF pain. This urine sample will be analysed for Complement activation products such as C3a and C5a. Diagnostic end points will be acquired through the routine management of these patients and accessed via the hospital imaging (PACS) and pathology (IHCS) reporting system. These will include appendix histology and microbiology, urinalysis, blood cultures, imaging and cervical swabs.

Table 1Blood Sample Assay Schedule Time Point Time of Test Routine Test Additional Trial Test Trial Assays Day Timings (example) PM Timings (example)

1. t = 0 Admission to A&E

   CONSENT ROUTINE:

   WCC, CRP, LFTs, Amylase, Clotting. Urinalysis.

   On attending clinicians discretion:

   urine culture, blood cultures, cervical swabs, imaging: US, CT, mri. Serum: C3, C4, C3dg, compliment activation markers

   Urine: compliment activation markers eg: C3a, C5a. 09:00 hrs 18:00 hrs
2. t = 1-4 h CONSENT(if not previously obtained) 09:00 to 13:00 hrs 1800 to 22:00 hrs
3. t = 4 h Trial Sample NO.1 C3, C4, C3dg,compliment activation markers 13:00 hrs 22:00 hrs
4. t =8h Trial Sample NO.2 C3, C4, C3dg, compliment activation markers 17:00hrs 02:00 hrs

   No action: 'blood taking curfew'
5. t = 12 h Trial Sample NO. 3 C3, C4, C3dg, compliment activation markers 21:00 hrs 06:00 hrs

   No action: 'blood taking curfew'
6. t = 23 h ROUTINE C3, C4, C3dg, compliment activation markers 08:00hrs t = 14 h 08:00 hrs
7. t = 47 h ROUTINE C3, C4, C3dg, compliment activation markers 08:00hrs t = 38 h 08:00 hrs
8. t = 71 h

   Some Patients Discharged

   Some patients for Laparoscopy ROUTINE C3, C4, C3dg, compliment activation markers 08:00hrs t = 62 h 08:00 hrs
9. If for surgery:

   t = surg0

   On Induction Trial Sample NO. 4 C3, C4, C3dg, compliment activation markers, CRP 09:00 hrs t = surg 0 21:00 hrs
10. t = surg 45 min

    End of surgery Pathology: appendix specimen Microbiology: appendix swabs Trial Sample NO. 5 C3, C4, C3dg, compliment activation markers, CRP 09:45 hrs t = surg 60 min 22: 00 hrs
11. t = x d, y h (days, hours from t0) Routine tests as they occur C3, C4, C3dg, compliment activation markers, CRP
12. Discharge

If readmitted within 14 days

tR=x d, y h(days, hours from t0) ROUTINE C3, C4, C3dg, compliment activation markers, CRP

The assays deployed for the CDAA pilot trial will include the current biomarkers of Complement consumption, C3 and C4, available in the clinical chemistry laboratory; in addition the investigators will use a panel of activation markers including C3dg, C4d, Bb and TCC that have been developed during the CPOP clinical trial. Prof Shaw's group now has extensive experience with the development, optimisation and internal auditing of the activation assays. The assay for the trial will be performed in Prof Shaw's laboratory in parallel with the clinical chemistry laboratory who will be responsible for producing aliquots from the plasma

ELIGIBILITY:
Inclusion Criteria:

* Admission for right iliac fossa pain

Exclusion Criteria:

Under 18 years unwilling to provide informed consent pregnant women diabetic immunosuppressed immunosuppression or steroid treatment within last 12 months learning disability Non-english speakers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 70 patients presenting with right Iliac Fosse pain
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2012-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Complement Activation differential diagnosis of Acute Appendicitis in a patient cohort presenting with Right Iliac Fosse Pain | up to 5 days
  C3 and C4 plasma concentration were measured in units of g/L over the time course t= admission, 4,8,12,23,47,71 hours or until discharge.
  Activation measures were derived as C3 and C4 differences at time each time point compared with admission values to derive changes in concentration which were compared in patients with a positive pathology diagnosis of the excised appendix (AA Group) and patients with a negative pathology diagnosis of the excised appendix or those patients discharged without appendectomy (non-AA Group).

SECONDARY OUTCOMES:
clinical Alvarado Score | up to 5 days
  The clinical Alvarado Score was derived for all patients on admission. Symptoms: Migration - score 1, Anorexia-acetone - score 1, Nausea-vomiting - score 1; Signs: Tenderness in the right lower quadrant - score 2, Rebound pain - score 1, Elevation in temperature - score 1; Laboratory: Leucocytosis - score 2, Shift to the left (i.e. neutrophils more than 75% of WCC) - score 1. Scores were compared in patients with a positive pathology diagnosis of the excised appendix (AA Group) and patients with a negative pathology diagnosis of the excised appendix or those patients discharged without appendectomy (non-AA Group).
The clinical Alvarado Score modified to include CRP > 5 mg/L - score 1 | up to 5 days
  The clinical Alvarado Score modified to include CRP > 5 mg/L - score 1and was derived for all patients on admission. Symptoms: Migration - score 1, Anorexia-acetone - score 1, Nausea-vomiting - score 1; Signs: Tenderness in the right lower quadrant - score 2, Rebound pain - score 1, Elevation in temperature - score 1; Laboratory: Leucocytosis - score 2, Shift to the left (i.e. neutrophils more than 75% of WCC) - score 1. Scores were compared in patients with a positive pathology diagnosis of the excised appendix (AA Group) and patients with a negative pathology diagnosis of the excised appendix or those patients discharged without appendectomy (non-AA Group).
Complement Activation Derived from C3dg | up to 5 days
  C3dg plasma concentrations were measured in units of micrograms/mL over the time course t= admission, 4,8,12,23,47,71 hours or until discharge.
  Activation measures were derived as C3 and C4 differences at time each time point compared with admission values to derive changes in concentration which were compared in patients with a positive pathology diagnosis of the excised appendix (AA Group) and patients with a negative pathology diagnosis of the excised appendix or those patients discharged without appendectomy (non-AA Group).
Complement Activation Terminal Cascade Complex | up to 5 days
  Terminal Cascade Complex plasma concentrations measured in units of ng/mL over the time course t= admission, 4,8,12,23,47,71 hours or until discharge.
  Activation measures were derived as C3 and C4 differences at time each time point compared with admission values to derive changes in concentration which were compared in patients with a positive pathology diagnosis of the excised appendix (AA Group) and patients with a negative pathology diagnosis of the excised appendix or those patients discharged without appendectomy (non-AA Group).
Complement Activation C3a in Urine | up to 5 days
  C3a concentrations in urine were measured in units of ng/mL over the time course t= admission, 4,8,12,23,47,71 hours or until discharge.
  Activation measures were derived as C3 and C4 differences at time each time point compared with admission values to derive changes in concentration which were compared in patients with a positive pathology diagnosis of the excised appendix (AA Group) and patients with a negative pathology diagnosis of the excised appendix or those patients discharged without appendectomy (non-AA Group).
C Reactive Protein Acute Phase Marker | up to 5 days
  C reactive protein serum concentrations were measured in units of mg/L over the time course t= admission, 4,8,12,23,47,71 hours or until discharge.
  Acute Phase measures were derived as C3 and C4 differences at time each time point compared with admission values to derive changes in concentration which were compared in patients with a positive pathology diagnosis of the excised appendix (AA Group) and patients with a negative pathology diagnosis of the excised appendix or those patients discharged without appendectomy (non-AA Group).

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Shaw, PhD, Principal Investigator — University of Exeter
Locations (1):
- Royal Devon & Exeter Foundation NHS Trust, Exeter, Devon, United Kingdom